CLINICAL TRIAL: NCT06803043
Title: A Randomized Controlled Trial to Evaluate a Trauma-Informed Partner Violence Intervention Program
Brief Title: Evaluation of a Trauma-Informed Partner Violence Intervention Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Rhode Island Hospital (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-45014; BPS-2023C1-31039 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Domestic Violence; Post Traumatic Stress Disorder
Keywords: Strength at Home (SAH); Group intervention; Motivational strategies; Justice-involved men; Alcohol use; Alexithymia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcohol Drinking; Affective Symptoms

STUDY DESIGN:
Intervention Model Description: A mixed-methods approach will be used for this single site, parallel group RCT. Participants will be randomized at the individual level to Strength at Home (SAH) or Treatment as Usual (TAU), with a 1:1 allocation ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength at Home (SAH) (Experimental): SAH isa trauma-informed 12-week intimate partner violence (IPV) intervention program.
  Interventions: Behavioral: SAH
- Treatment as Usual (TAU) (Active Comparator): TAU is a 20-week state-approved IPV intervention program.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: SAH — SAH is a group trauma informed intervention that uses motivational strategies and self-monitoring of one's thoughts and responses. It provides a unique fusion of interventions for trauma and IPV and consists of 12 two-hour weekly sessions. Throughout the program, group members complete in-session practice exercises and are provided "practice assignments" to consolidate and apply information learned in group.
  Arms: Strength at Home (SAH)
Behavioral: TAU — TAU is a court mandated 20 week, psychoeducational/directed program that emphasizes the sharing of power and control in relationships and personal accountability. Topics also focus on equality wheels, substance abuse impacts, culture and socialization impact on gender roles, defense mechanisms versus coping skills, triggers for stress and anger, and healthy versus unhealthy communication.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this study is to conduct a randomized controlled trial (RCT) comparing outcomes between two programs to reduce intimate partner violence (IPV)- the Strength at Home (SAH) program and a standard, state-approved IPV intervention program, Treatment as Usual (TAU). Primary outcomes will include self- and partner-reported physical and psychological IPV. Secondary outcomes will include self-reported PTSD symptoms, alexithymia, alcohol use problems, and treatment satisfaction, assessed across five time points.

DETAILED DESCRIPTION:
A mixed-methods approach will be used for this single site, parallel group RCT. All participants will be randomized at the individual level to Strength at Home (SAH) or Treatment as Usual (TAU), with a 1:1 allocation ratio. Assessments will occur pre-treatment and post-treatment with follow-up assessments scheduled every three months post-treatment through month 12. Assessments have been designed to examine reductions in IPV and other outcomes including posttraumatic stress disorder (PTSD) symptoms and alcohol use.

The primary hypotheses are that those receiving SAH will evidence greater reductions in physical and psychological IPV, symptoms of PTSD, alexithymia, and alcohol use problems, and higher treatment satisfaction relative to those receiving TAU across the time points.

The specific aims and sub aims are:

1. Test the comparative effectiveness of SAH and TAU by conducting an RCT comparing 200 justice-involved men randomly assigned to each program.

   * Compare the frequency of physical and psychological IPV, the primary outcomes of interest, across conditions as reported by the male participants and their intimate partners across Time 1 (baseline) and four 3-month follow ups (Times 2-5). Additionally, at Time 5, the study may make use of available arrest record data from the state of Rhode Island.
   * Compare symptoms of PTSD, alexithymia, and alcohol use problems across conditions and assessment time points as reported by the male participants.
   * Compare treatment satisfaction across conditions as reported by the male participants across the four 3-month follow ups (Times 2-5).
2. Facilitate future use of SAH by working closely with the Stakeholder Advisory Board to identify potential barriers and facilitators to successful implementation in civilian community settings.

   * Identify barriers and facilitators to implementation.
   * Assess the acceptability of SAH among stakeholders in the community setting and areas in need of refinement.

ELIGIBILITY:
Inclusion Criteria:

* Men court-mandated to IPV intervention from the Rhode Island Department of Parole and Probation and their partners

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
IPV Assessment | Baseline, 3 months, 6 months, 9 months, 12 months
  The Revised Conflict Tactics Scale (CTS2) is a 39-item measure of individual engagement in or experience of physical or psychological violence with an intimate partner. Each item is asked about both the respondent and the respondent's partner, for a total of 78 questions.The response options include 8 choices (Categories 1-7 and 0). An answer of Category 1 or 2 is coded as the corresponding number of times the specified incident occurred (once or twice in the past year). For Categories 3-5, the midpoint of the category is coded. For example: Category 3 (3-5 times) is coded as 4, Category 4 (6-10 times) is coded as 8, and Category 5 (11-20 times) is coded as 15. Category 6 (More than 20 times) should be coded as 25. Category 7 is given a score of 0 if scores for the previous year do not reflect abuse or conflict. Total scores can range from 0 to 975 and lower scores suggest less conflict.
Psychological IPV Assessment | Baseline, 3 months, 6 months, 9 months, 12 months
  The 7-item Restrictive Engulfment subscale of the Multidimensional Measure of Emotional Abuse (MMEA) will be used as an additional measure of psychological IPV. Each item has 7 potential responses from 0=never to 6= more than 20 times. Scores can range from 0 to 42, with higher scores being associated with more psychological IPV.

SECONDARY OUTCOMES:
Post traumatic stress disorder (PTSD) | Baseline, 3 months, 6 months, 9 months, 12 months
  The 20-item PTSD Checklist for DSM 5 (PCL-5) will be used to assess PTSD symptoms. It is a self-report measure. Items are rated on a 5-point Likert scale [0 to 4] and summed. Scores range from 0 to 80 with higher scores associated with more PTSD symptoms. A total score of 33 or higher may indicate severe PTSD.
Alexithymia | Baseline, 3 months, 6 months, 9 months, 12 months
  The 20-itemToronto Alexithymia Scale (TAS-20) will be used to assess alexithymia. The TAS-20 uses cutoff scoring, with scores of 52-60 indicating possible alexithymia, and scores above 60 indicating alexithymia.
Alcohol Use | Baseline, 3 months, 6 months, 9 months, 12 months
  Alcohol use will be assessed by the Alcohol Use Disorders Identification Test (AUDIT). AUDIT has 10 questions and the possible responses to each question are scored 0, 1, 2, 3 or 4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol.
Treatment satisfaction | 3 months, 6 months, 9 months, 12 months
  Participants' satisfaction will be assessed with a 4-item measure used in a study conducted by the Treatment of Depression Collaborative Research Program.

CONTACTS AND LOCATIONS:
Overall Officials: Casey T Taft, PhD, Principal Investigator — CABU School Medicine, Psychiatry; Lindsay Orchowski, PhD, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - CABU School of Medicine, Psychiatry, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No